CLINICAL TRIAL: NCT06861803
Title: Comparison of Laboratory and Ultrasound Findings Between Letrozole-Resistant and Letrozole-Sensitive PCOS Patients in Egypt
Brief Title: Laboratory and Ultrasound Findings and Response to Letrozole in PCOS Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, lecturer and consultant at Obstetrics and Gynecology Department., Al-Azhar University
Other Study IDs: Gyne19225
Record Dates: First submitted 2025-02-18; First posted 2025-03-06 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: PCOS (Polycystic Ovary Syndrome) of Bilateral Ovaries
Keywords: PCOS; letrozole
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PCOS patients: The study will include a single group of women diagnosed with polycystic ovary syndrome (PCOS) based on the Rotterdam criteria, who are undergoing ovulation induction with letrozole for the first time. Participants will be women aged 18-40 years attending the outpatient clinic at Al-Hussein University Hospital for infertility treatment. All participants will undergo a comprehensive baseline assessment, including clinical evaluation, laboratory investigations, and transvaginal ultrasound before starting letrozole therapy. After treatment, they will be classified into letrozole-sensitive or letrozole-resistant subgroups based on their ovulatory response. The study aims to identify potential predictors of letrozole resistance by comparing baseline characteristics between these two outcome-based subgroups.
  Interventions: Drug: Letrozole tablets

INTERVENTIONS:
Drug: Letrozole tablets — The intervention in this study is ovulation induction using letrozole, an aromatase inhibitor commonly used in women with polycystic ovary syndrome (PCOS) to stimulate ovulation. Participants will receive letrozole at an initial dose of 2.5 mg/day for five days, starting on day 3 of the menstrual cycle. If ovulation is not achieved, the dose will be incrementally increased up to a maximum of 7.5 mg/day over a maximum of three cycles. Ovulation will be monitored through serial transvaginal ultrasounds to assess follicular development, and confirmed by measuring mid-luteal serum progesterone levels (>3 ng/mL). Based on the response to letrozole, participants will be classified as either letrozole-sensitive (ovulatory) or letrozole-resistant (anovulatory) to identify potential predictors of resistance and improve individualized treatment strategies for PCOS-related infertility.

SUMMARY:
The goal of this observational study is to compare laboratory and ultrasound findings between letrozole-resistant and letrozole-sensitive PCOS patients in Egypt. The study will include women aged 18-40 years diagnosed with PCOS based on the Rotterdam criteria, who are undergoing ovulation induction with letrozole for the first time.

The main questions it aims to answer are:

What are the baseline laboratory and ultrasound differences between letrozole-resistant and letrozole-sensitive PCOS patients? What factors can predict letrozole resistance in PCOS patients? Researchers will compare letrozole-resistant and letrozole-sensitive PCOS patients to determine whether specific laboratory markers and ultrasound findings can predict resistance to letrozole.

Participants will:

Undergo baseline clinical, laboratory, and ultrasound assessments before starting letrozole treatment.

Receive letrozole treatment with dose escalation up to 7.5 mg/day over a maximum of three cycles if ovulation is not achieved.

Be monitored through serial transvaginal ultrasounds to assess follicular development.

Have ovulation confirmed via mid-luteal serum progesterone levels. The study aims to improve the understanding of predictors of letrozole resistance to guide personalized ovulation induction strategies in PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-40 years.
* Diagnosis of PCOS based on Rotterdam criteria.
* No prior ovulation induction with letrozole.
* Willing to follow the treatment protocol and attend follow-up visits

Exclusion Criteria:

* Infertility due to other causes such as tubal obstruction or male factor infertility.
* Previous ovarian surgery or use of medications that could influence ovulation.
* Comorbidities such as uncontrolled diabetes, hyperprolactinemia, or thyroid dysfunction.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study will include female participants only, as it focuses on women diagnosed with polycystic ovary syndrome (PCOS) who are undergoing ovulation induction with letrozole for infertility treatment. Male participants are not eligible for this study.
Study Population: The study will include women diagnosed with polycystic ovary syndrome (PCOS) based on the Rotterdam criteria, who are seeking infertility treatment and undergoing ovulation induction with letrozole for the first time. Participants will be women aged 18-40 years, recruited from the outpatient clinic at Al-Hussein University Hospital, a tertiary healthcare center in Egypt. All participants will undergo a comprehensive baseline assessment, including clinical evaluation, laboratory investigations, and transvaginal ultrasound before starting letrozole treatment. The study aims to identify potential predictors of letrozole resistance by comparing baseline characteristics between women who respond to treatment and those who do not.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of baseline FSH level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline FSH level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline LH level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline LH level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline LH/FSH ratio level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline LH/FSH ratio level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline AMH level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline AMH level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline total testosterone level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline total testosterone level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline fasting insulin level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline fasting insulin level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline glucose level between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline glucose level between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline lipid profile between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days).
  This outcome measures the differences in baseline lipid profile between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline antral follicle count between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days)
  This outcome measures the differences in baseline antral follicle count between letrozole-sensitive and letrozole-resistant PCOS patients.
Comparison of baseline ovarian volume between letrozole-sensitive and letrozole-resistant PCOS patients. | At the end of cycle 3 of treatment (each cycle is 28 days)
  This outcome measures the differences in baseline ovarian volume between letrozole-sensitive and letrozole-resistant PCOS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muhamed Alhagrasy, M.D., Principal Investigator — Al-Azhar University
Locations (1):
- Al-Hussein University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study investigators will share de-identified individual participant data (IPD) related to baseline laboratory and ultrasound findings, ovulation outcomes, and relevant clinical parameters. The shared dataset will exclude any personally identifiable information to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available six months after study completion and will remain accessible for a period of five years.
Access Criteria: Researchers and qualified investigators may request access to the dataset for scientific and academic purposes. Requests must be submitted to the corresponding author via email and include a research proposal outlining the intended use of the data. Access will be granted upon approval by the study team, and data users must agree to a data use agreement ensuring confidentiality and ethical use of the shared information.